CLINICAL TRIAL: NCT03078023
Title: Is EPO Staining on Esophageal Sponge Samples a Simple Reliable Method of Accessing Esophageal Eosinophilia?
Brief Title: Sponge and Eosinophil Peroxidase (EPO) Staining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karthik Ravi, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-009403
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Toothbrushing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- swallowed sponge device (Experimental): Swallowing a sponge prior to a clinical upper endoscopy. Patients diagnosed with Eosinophilic Esophagitis (EoE) > than 15 Eosinophils per high power field (phf) and failed to respond to Proton Pump Inhibitors (PPI) therapy. Will be asked to swallow a sponge, this is a 10 minute procedure done in the office prior to their clinical upper endoscopy. This will be sent for histology, >15 Eos phf would be considered active disease. We will compare the results of the sponge using the EPO staining technique compared to histologic response.
  Interventions: Device: swallowed sponge device

INTERVENTIONS:
Device: swallowed sponge device — Swallowed sponge: Subjects having a clinical upper endoscopy will be asked to swallow the sponge 2 hours prior to EGD
  Other Names: brush

SUMMARY:
Are we able to use the EPO staining technique using the sponge ?

DETAILED DESCRIPTION:
EPO staining on esophageal sponge samples had a strong association with peak esophageal eosinophil counts on endoscopic biopsy specimens in a small study of 26 patients Using a cut-off of 1.1 absorbance units in a colorimetric assay at a wavelength of 492nm the EPO stain had sensitivity and specificity of 1105 and 83% respectively for a peak eosinophil count of 15 eos/hpf on histologic endoscopic obtained biopsy specimens. The technique of EPO staining is standardized and can be completed in 45 minutes time. Currently, we have found esophageal sponge cytology sensitive and specific for assessment of esophageal eosinophilia. It allows disease activity assessment without endoscopy is much preferred by patients over the standard endoscopic technique of disease assessment. The process of specimen preparation in fairly tedious and interpretation takes significant experience. If EPO staining on non-endoscopic esophageal sponge studies was accurate at assessing disease activity, this is a tool that could be easily performed and interpreted with a rapid turnaround time.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Diagnosed with Eosinophilic Esophagitis > than 15 Eos phf and failed to respond to the PPI therapy
* Going through the six food elimination diet or have just completed elimination the six foods: fish, nuts, eggs, soy, wheat, and milk

Exclusion Criteria:

* Clinical evidence of infectious process potentially contributing to dysphagia (e.g. candidiasis, CMV, herpes)
* Other cause of dysphagia identified at endoscopy (e.g. reflux esophagitis, stricture, web, ring, achalasia, esophageal neoplasm)
* Esophageal minimal diameter < 13 mm on structured barium esophagram

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Sponge pathology verses biopsy results: number of eosinophils | 1 year
  Patients will swallow the sponge prior to a clinical upper endoscopy with biopsies. We will compare upper endoscopy biopsies to the pathology from the cytosponge using the EPO staining technique.

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ravi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials